CLINICAL TRIAL: NCT04728412
Title: High Flow Oxygen Therapy in Patients With or at Risk of Respiratory Failure Undergoing Felxible Bronchoscopy Under Sedation: a Pilot Study
Brief Title: High Flow Oxygen Therapy in Patients Undergoing Bronchoscopy Under Sedation
Acronym: BroncHoFlow
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardarelli Hospital (Other)
Responsible Party: Principal Investigator, Giuseppe Failla, Chief of Interventional Pulmonology Unit, Cardarelli Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00000
Record Dates: First submitted 2020-12-12; First posted 2021-01-28 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Failure; Hypercapnic Acidosis
Keywords: bronchoscopy; sedation; high flow oxygen therapy
MeSH Terms: conditions — Respiratory Insufficiency; Acidosis, Respiratory

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients undergoing bronchoscopy under sedation with or at risk of respiratory failure (Experimental)
  Interventions: Device: High Flow Oxygen Therapy (HFOT)

INTERVENTIONS:
Device: High Flow Oxygen Therapy (HFOT) — HFOT administration in patients undergoing bronchoscopy under moderate sedation, affected by or at risk of hypoxemic and/or hypercapnic respiratory failure.

SUMMARY:
A reduction of peripheral oxygen saturation (SpO2) commonly occurs during bronchoscopy and may be associated with both respiratory and cardiac adverse events. The type of breathing assistance that should be delivered to patients, in order to treat and/or to prevent acute respiratory failure, during or after bronchoscopy, is not universally standardized; studies comparing the impact of different respiratory supports on patient's outcome and on hospital resource use are very few. the risk of respiratory failure rises according to the type of procedure (i.e., increased risk with broncho-alveolar lavage and trans-bronchial lung biopsy) and to the use of sedative drugs. Conventional oxygen therapy with nasal cannula, continuous positive airway pressure and non-invasive ventilation are commonly applied during endoscopic procedures. High flow oxygen therapy (HFOT) is a relatively novel device, still under-used in the context of interventional pulmonology, providing an humidified air-oxygen blend up to 60 L/min. HFOT has been reported to be effective for the treatment of both hypoxemic and hypercapnic respiratory failure. The investigators hypothesize that HFOT could be feasible and safe in patients undergoing bronchoscopy under moderate sedation, affected by or at risk of hypoxemic and/or hypercapnic respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* pH ≥7.30 e PaCO2 >45 mmHg and/or
* PaO2/FiO2 <300 mmHg o SpO2 <90 percent on room air
* Patient at risk of respiratory failure (COPD III-IV GOLD stage; OSAS; restrictive lung and chest wall diseases; cardiac failure)

Exclusion Criteria:

* Need of laryngeal mask and/or
* Patients on NIV for >16 hrs/day and/or
* pH <7.30 and/or
* Tracheostomy and/or
* Recent (<3 months) facial trauma and/or
* Hemodynamic instability and/or
* High risk of aspiration and/or
* Lacerated trachea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of desaturation, defined as SpO2< 90 percent percent for >1 min, <5. | one year
Percent of variation of pH, comparing ABG performed before bronchoscopy with that performed before partecipant's transferral to recovery room. | one year
Percent of variation of PaCO2 variation, comparing ABG performed before bronchoscopy with that performed before partecipant's transferral to recovery room. | one year
Rate of interruption of bronchoscopy because of number of desaturation, defined as SpO2< 90 percent for >1 min, >5. | one year
Number of partecipants requiring an escalation of respiratory support. | one year
Rate of new appearance of hemodynamic instability. | one year

SECONDARY OUTCOMES:
value of Charlson Comobidity Index associated with HFOT failure. | one year
value of Body Mass Index associated with HFOT failure. | one year
value of Borg dyspnea scale associated with HFOT failure. | one year
Number of desaturations, defined as SpO2< 90 percent for >1 min. | one year
Lowest oxygen saturation under HFOT. | one year
Rate of change of HFOT parameters because of desaturation without respiratory acidosis. | one year
Rate of change of HFOT parameters because of desaturation with respiratory acidosis | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Giuseppe Failla, MD, Naples, Italy